CLINICAL TRIAL: NCT00581204
Title: Development of an Algorithm for Prediction of Onset of Hemodynamic Instability in Humans
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Brooke Army Medical Center (U.S. Federal Agency); Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Matthew Brenner, M.D.,Department of Pulmonary and Critical Care Medicine, University of California, Irvine
Other Study IDs: 20065191
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Hemorrhagic Shock
Keywords: trauma situations; Lower Body Negative Pressure (LBNP)
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Tool: Near-Infrared Diffuse Optical Spectroscopy Imaging
  Interventions: Device: Near-Infrared Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Near-Infrared Diffuse Optical Spectroscopy — Early predictor of hemorrhagic shock
  Other Names: Near-Infrared Diffuse Optical Spectroscopy Imaging

SUMMARY:
The purpose for this study is to measure the physiology of human undergoing a Lower Body Negative Pressure usea non-invasive low-power optical technique, near-infrared diffuse optical spectroscopy measurement and compare these measurement to standard monitoring procedures delineated in the Brooke Army Medical Center.

The Brooke Army Medical Center can use near-infrared diffuse optical spectroscopy to provide functional physiologic tissue and organ information without ionizing radiation and without withdrawing any blood, in a cost-effective and rapid manner. Monitoring for the onset of circulatory shock in a wounded soldier on the battlefield is typically performed by measurement of arterial blood pressure, arterial oxygen saturation, or simple auscultation of the pulse. Shock is typically recognized by non-specific signs and subjective symptoms such as cold clammy skin, pallor, weak thready pulse, unstable vital signs, and diminished mentation.

DETAILED DESCRIPTION:
The near-infrared diffuse optical spectroscopy can measure tissue regions deeper below the skin surface and reports on larger tissue volumes in muscle and brain. The near-infrared diffuse optical spectroscopy instrument generate harmless amounts of low-level non-ionizing near-infrared ligh can measure the tissue absorption and scattering properties at depths of 1 cm or more below the skin surface include larger tissue volumes in muscle and brain. The absorption properties of tissue provide and can determine absolute concentrations of deoxygenated hemoglobin, oxygenated hemoglobin, and water, as well as the total hemoglobin saturation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy nonsmoking normotensive males or females.
* Age 18 to 55 years old, Military or civilian.
* Active duty military members who are 17 years old

Exclusion Criteria:

* Age <18 and >55 years, except for 17 year old active duty military members.
* History of hyperthyroidism,hypertension, cardiovascular abnormalitY, respiratory illnesses,anaphylaxis,pre-syncopal/syncopal episodes,abnormal blood clotting,
* Taking drugs to alter autonomic function
* History of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Army Medical Center, civilian and military
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Early predictor of shock | 5 to 60 seconds.
  The near-infrared diffuse optical spectroscopy measure tissues properties

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brenner, M.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute,University of California, Irvine, Irvine, California, United States